CLINICAL TRIAL: NCT00946946
Title: Double-blind, Double-dummy, Randomised, Multicentre, Comparative Study on the Efficacy and Safety of Azathioprine Versus Mesalazine for Prevention of Clinical Relapses in Crohn's Disease Patients With Postoperative Moderate or Severe Endoscopic Recurrence
Brief Title: Preventing Postoperative Relapse in Crohn's Disease Patients at Risk: Azathioprine Versus Mesalazine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AZT-2/CDP
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Crohn's Disease
Keywords: Randomized; Crohn's Disease; Prevention; Azathioprine; mesalazine; mesalamine; TPMT
MeSH Terms: conditions — Crohn Disease | interventions — Azathioprine; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azathioprine (Experimental): 2.0-2.5 mg/kg/BW azathioprine tablets/day AND mesalazine placebo tablets
  Interventions: Drug: Azathioprine; Drug: Mesalazine placebo
- Mesalazine (Active Comparator): 4g mesalazine tablets/day AND azathioprine placebo tablets
  Interventions: Drug: Mesalazine; Drug: Azathioprine placebo

INTERVENTIONS:
Drug: Azathioprine — 2.0-2.5mg/kg/BW azathioprine /day and mesalazine placebo tablets
  Other Names: Azafalk 50mg tablets
  Arms: Azathioprine
Drug: Mesalazine — 4g Mesalazine tablets/day AND azathioprine placebo tablets
  Other Names: Salofalk 500mg tablets
  Arms: Mesalazine
Drug: Azathioprine placebo — 4g Mesalazine tablets/day AND azathioprine placebo tablets
  Arms: Mesalazine
Drug: Mesalazine placebo — 2.0-2.5mg/kg/BW azathioprine /day and mesalazine placebo tablets
  Arms: Azathioprine

SUMMARY:
This study aims to compare azathioprine versus mesalazine tablets for the prevention of clinical relapse in postoperative Crohn's disease (CD) patients with moderate or severe endoscopic recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Man or woman between 18 and 70 years of age,
* Diagnosis of Crohn's disease confirmed by endoscopic and histological, or endoscopic and radiological criteria within one year or by histopathological criteria during resection,
* Clinical remission defined as Crohn´s Disease Activity Index (CDAI) < 200, within the last two weeks. No clinical relapse due to Crohn's disease since resection,
* Moderate (i2a) or severe endoscopic recurrence (i3-i4) within 6 to 24 months after curative resection of the terminal ileum and partial colectomy with ileocolonic resection for complications of ileal Crohn´s disease and with a construction of an ileocolonic anastomosis,
* Within the neoterminal ileum at least more than 5 aphthous lesions with normal mucosa between the lesions, or skip areas of larger lesions,
* Negative pregnancy test at screening visit in females of childbearing potential,
* Use of appropriate contraceptive methods for females of childbearing potential and males with procreative capacity during treatment and at least up to 3 months after the end of treatment.

Exclusion Criteria:

* Lesions confined to the ileocolonic anastomosis (i.e., < 1 cm in length)
* Short bowel syndrome,
* Serious secondary illnesses of an acute or chronic nature, which in the opinion of the Investigator renders the patient unsuitable for inclusion into the study,
* Serum creatinine levels exceeding 1.5 mg/dL or 130 umol/L,
* Presence of an ileo-/colonic stoma,
* Genotype: thiopurine methyltransferase (TPMT) -/-,
* Known previous or concurrent malignancy (other than that considered surgically cured, with no evidence for recurrence for 5 years),
* Treatment with cytostatics or immunosuppressants, methotrexate, cyclosporine, 6-MP, Azathioprine, 6-TG or anti-TFN-alpha therapy since resection; postoperative treatment with corticosteroids for more than 4 weeks or postoperative treatment with oral antibiotics (e.g., metronidazole, ciprofloxacin) for more than 4 weeks,
* Application of non-steroidal anti-inflammatory drugs (NSAIDS) within 2 weeks before Screening visit except low dose acetylsalicylic acid and except paracetamol,
* Known intolerance/hypersensitivity to study drugs or drugs of similar chemical structure or pharmacological profile,
* Scheduled or intended active immunisation with living vaccines within the next 12 months,
* Well-founded doubt about the patient's cooperation,
* Existing pregnancy, lactation, or intended pregnancy or impregnation within the next 15 months,
* Non-use of appropriate contraceptives in males with procreative capacity and females of childbearing potential (e.g. condoms for males, intrauterine device [IUD], hormonal contraception for females, or a means of contraception for a particular patient considered adequate by the responsible investigator) during treatment and within 3 months after the end of treatment,
* Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial,
* Present stricture plasty (no exclusion if the present stricture plasty was macroscopically without any relevant finding of inflammation seen during index surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2002-02; Primary Completion 2007-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was therapeutic failure at one year, defined as CDAI score ≥200 and an increase of ≥60 points from baseline, or study drug discontinuation due to lack of efficacy or intolerable adverse drug reaction. | 12 months

SECONDARY OUTCOMES:
endoscopic improvement at month 12, defined as ≥1 point reduction in Rutgeerts' score. | 12 months
change in CDAI score | 12 months
adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Walter Reinisch, Prof, Principal Investigator — Universitaetsklinik für Innere Medizin III, Abteilung Gastroenterologie and Hepatologie, Vienna, Austria
Locations (2):
- Universitaetsklinik für Innere Medizin III, Abteilung Gastroenterologie and Hepatologie, Vienna, Austria
- Robert-Bosch Krankenhaus, Innere Medizin I, Stuttgart, Germany

REFERENCES:
- [Result] Reinisch W, Angelberger S, Petritsch W, Shonova O, Lukas M, Bar-Meir S, Teml A, Schaeffeler E, Schwab M, Dilger K, Greinwald R, Mueller R, Stange EF, Herrlinger KR; International AZT-2 Study Group. Azathioprine versus mesalazine for prevention of postoperative clinical recurrence in patients with Crohn's disease with endoscopic recurrence: efficacy and safety results of a randomised, double-blind, double-dummy, multicentre trial. Gut. 2010 Jun;59(6):752-9. doi: 10.1136/gut.2009.194159. PMID 20551460